CLINICAL TRIAL: NCT06795932
Title: Prise En Charge Des Atteintes Proprioceptives Chez Une Population Avec Capsulite Rétractile
Brief Title: Evaluation and Treatment of Adhesive Capsulitis Using Non-invasive Neurostimulation Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-UQAC : 2025-1773
Record Dates: First submitted 2024-11-14; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-11

CONDITIONS: Adhesive Capsulitis of the Shoulder; Frozen Shoulder
Keywords: Adhesive Capsulitis; Frozen shoulder; Tendon Vibration; Transcranial Magnetique Stimulation; Proprioception; Kinesthetic illusions
MeSH Terms: conditions — Bursitis; Illusions

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tendon vibration and standardized exercise protocol (Experimental): Six interventions inducing kinesthetic illusions (20 minutes, 1 illusion/minute).
  Two interventions per week, for three weeks. Accompanied by a daily exercise protocol.
  Interventions: Device: Tendon Vibration; Other: Exercices
- Tendon vibration without kinesthetic illusion and standardized exercise protocol (Sham Comparator): Six interventions not inducing kinesthetic illusions (20 minutes) Two interventions per week, for three weeks. Accompanied by a daily exercise protocol.
  Interventions: Other: Exercices; Device: Tendon vibration

INTERVENTIONS:
Device: Tendon Vibration — Vibration can create kinesthetic illusions when applied at some modalities. The vibration will be put at 80 Hz and 1 mm of amplitude for 10 seconds to create 1 illusion/minute, during 20 minutes.
  Two interventions per week, for three weeks. Total : 6 interventions
  Arms: Tendon vibration and standardized exercise protocol
Other: Exercices — Standardized exercise protocol, performed daily for 3 weeks, with a diary.
Device: Tendon vibration — Tendon vibration will not induce kinesthetic illusions, since it will be applied 40 Hz and 1 mm of amplitude for 10 seconds.
  Two interventions per week, for three weeks. Total : 6 interventions
  Arms: Tendon vibration without kinesthetic illusion and standardized exercise protocol

SUMMARY:
The goal of this randomized controlled trial is to compare the integrity of somatosensory processing with transcranial magnetique stimulation (TMS) and corticospinal excitability of the affected shoulder in individuals with adhesive capsulitis versus healthy controls.

The secondary objective is to compare the clinical and neurophysiological effects of an intervention using tendon vibration (VIB) to induced kinesthetic illusions. This will involve comparing two groups: one receiving a real intervention versus a placebo intervention protocol, both coupled with standardized exercises in individuals with capsulitis. The hypotheses are that the proprioceptive processing and corticospinal excitability are impaired in the presence of capsulitis, and that the VIB + exercises intervention will result in greater improvements than the placebo VIB + exercises.

To goal is to establish the first empirical foundations for understanding adhesive capsulitis, using cutting-edge neurophysiological investigation technologies.

TMS will be used to explore the presence of maladaptive plasticity in motor networks by assessing the excitability and integrity of the primary motor cortex (M1) and the corticospinal tract.

Recruitement:

30 healthy participants and 30 participants with a diagnosis of adhesive capsulitis will undergo 2 baselines assesments, 6 interventions with tendon vibration and 2 follow-up evaluation. Participants will be age- and sex-matched.

Baseline and follw-up include:

* Questionnaires : SPADI, QuickDASH, French version of the Mcgill Pain Questionnaire;
* Active and passive range of motion;
* Ultrasound for diagnosing capsulitis.

Comparison parameters:

* active motor threshold (aMT)
* Motor evoked potential (MEP) latency and amplitude
* Standardized kinesthetic illusion procedure (SKIP) : direction of illusion, clearness, amplitude/speed.

Interventions :

* 2 baselines including all questionnaires, ultrasound, active and passive range of motion, TMS procedure and SKIP;
* 2 VIB interventions per week, for 3 weeks

  * Real VIB : 80Hz of vibration to induce kinesthetic illusions,
  * Placebo VIB : 40Hz of vibration that does not induce kinesthetic illusions
* 2 follow-up including all questionnaires, ultrasound, active and passive range of motion, TMS procedure and SKIP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Good general health
* Adhesive capsulitis (experimental group) or
* No shoulder pain (placebo group)

Exclusion Criteria:

* Cognitive disorders;
* Any neurological disease/injury affecting the upper limbs;
* History or diagnosis of muscle, tendon, or capsular tear;
* Shoulder surgery/prosthesis;
* Pregnant woman;
* Presence of metal in the skull or jaw;
* History of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And Disability Index | at baseline 1 and follow-up 1 : 2 months
  SPADI : Shoulder Pain And Disability Index Thirteen questions to quantify the level of difficulty, ranging from 0 to 10, based on pain and disability.
  Five questions assess pain (0 = no pain, 10= worst pain imaginable) and eight questions assess the level of difficulty in performing different tasks (0= no difficulty, 10=too difficult, need help).
Quick Disability of the Hand, Arm and Shoulder | at baseline 1 and follow-up 1: 2 months
  QuickDASH : Quick Disability of the Hand, Arm and Shoulder Allowing the calculation of a percentage ratio from 14 questions, using a visual analogue scale from 1 (no difficulty) to 5 (incapacity), on the effects of pain on daily life activities, work, and sports, in addition to associated symptoms such as paresthesia and sleep disturbances.
Questionnaire St-Antoine | at baseline 1 and follow-up 1: 2 months
  French version of McGill Pain Questionnaire. Subjectively assess the pain level with 16 questions on a scale from 0 (none) to 4 (extremely severe).
Range of motion | at baseline 1 and follow-up 1: 2 months
  Measuring the active and passive range of motion with a goniometer.
Standardized Kinesthetic Illusion Procedure | at baseline 1/2 and follow-up 1/2 : 2 months (+/- 2 weeks)
  Using the SKIP to evaluate:
  * Clarity: 0 = no illusion, 1 = vague, 2 = moderately clear, 3 = perfectly clear
  * Direction: using words
  * Speed/amplitude of illusion: using a visual analogue scale where participants mark a point on the line to represent the speed/amplitude (ranging between very slow/small to very fast/high)
Active motor threshold | at baseline 1-2 and follow-up 1-2: 2 months (+/- 2 weeks)
  The active motor threshold represents the intensity of stimulation (%) required to elicit measurable motor evoked potentials.
Amplitude of motor evoked potential | at baseline 1-2 and follow-up 1-2: 2 months (+/- 2 weeks)
  The measurement of the motor evoked potential amplitude (peak-to-peak) It corresponds to the amount of neurons stimulated at the central et peripheral levels, expressed in microvolts.
Latency of motor evoked potential | at baseline 1-2 and follow-up 1-2: 2 months (+/- 2 weeks)
  The measurement of the motor evoked potential latency in miliseconds. It represent the conduction time from the application of the stimuli over the cortex to the target muscle.

SECONDARY OUTCOMES:
Sociodemographic - age | at baseline 1 : 1 day
  Age of each participant, in months
Sociodemographic - Sex | at baseline 1: 1 day
  Physiological sex
Sociodemographic - Weight | at baseline 1: 1 day
  kilograms
Sociodemographic - Height | at baseline 1: 1 day
  in meters

CONTACTS AND LOCATIONS:
Locations (1):
- Lab BioNR - UQAC, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided